CLINICAL TRIAL: NCT04931277
Title: Stepped Surgery in Uveitic Cataract: A Novel Approach to a Quiet Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amgad Mahmoud El Nokrashy, Lecturer of Ophthalmology, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.21.01.1176
Record Dates: First submitted 2021-06-12; First posted 2021-06-18 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Outcome of Stepped Cataract Surgery in Uveitis
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stepped cataract surgery (Other)
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — stepped surgery in the form of primary phacoemulsification and secondary posterior chamber intraocular lens (PCIOL) implantation in patients with uveitis.

SUMMARY:
This study aims to assess the short-term results of primary phacoemulsification and secondary posterior chamber intraocular lens (PCIOL) implantation in patients with uveitis.

ELIGIBILITY:
Inclusion Criteria:

* the study will include any uveitic patients below 45 years old with complicated cataract and their best corrected visual acuity (BCVA) not better than 6/36 nor worse than hand movement

Exclusion Criteria:

* the study will not include those with visual acuity more than 6/36 or patients with active uveitis or with posterior segment pathology discovered by ultrasonography that may affect to a lager extent the visual prognosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Visulal acuity | 6 months
  overall improvement in vision using LogMAR

SECONDARY OUTCOMES:
Intraocular inflammation | 6 months
  flare up of inflammation after surgery USING SUN classification

CONTACTS AND LOCATIONS:
Overall Officials: Amgad El Nokrashy, MD, Principal Investigator — Mansoura University; Dina Abd El Fattah, MD, Study Chair — Mansoura University; Rania Bassiouny, MD, Study Chair — Mansoura University; Shreen Gaafar, MD, Study Chair — Mansoura University; Waleed Gaafar, MD, Study Director — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Dakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No
results